CLINICAL TRIAL: NCT00716118
Title: Oocytes Cryopreservation: The Impact of Cryopreservation on the Meiotic Spindle and Mitochondria of Human Oocytes.
Brief Title: Oocyte Cryopreservation: The Impact of Cryopreservation on the Meiotic Spindle and Mitochondria of Human Oocytes.
Acronym: WCFC
Status: Completed | Type: Observational
Sponsor: West Coast Fertility Centers (Other)
Responsible Party: David G. Diaz MD, West Coast Fertility Centers
Other Study IDs: 2008-02
Record Dates: First submitted 2008-07-11; First posted 2008-07-16 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Infertility
Keywords: Oocyte Cryopreservation; Slow-Freeze; Egg Freezing; Meiotic Spindle; Mitochondria; Human Oocytes Freezing.
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: IVF patients.

SUMMARY:
Our aims is to document the possible effect of cryo- preservation at the meiotic spindle and mitochondrial levels.

DETAILED DESCRIPTION:
The cryopreservation of oocytes (OC) has broad applications in the field of reproductive endocrinology for the management of clinical problems in both fertile and infertile patients. For example, young fertile women who are diagnosed with malignancies may freeze their oocytes before initiating potentially toxic radiation or chemical cancer therapy which may render them sterile.

Using the OC technology, we have established a frozen oocyte bank using healthy, compensated egg donors who have been pre- screened using FDA criteria. Following an appropriate quarantine time, oocytes can be thawed and offered to women diagnosed with premature ovarian failure or diminished ovarian reserve. This application of OC has already shown promise by eliminating the logistical and clinical complications associated with traditional oocyte donation using fresh oocytes from donors.

From the societal perspective, cryopreservation of surplus oocytes in an IVF cycle may remove some of the social and moral objections surrounding embryo cryopreservation. Currently, our frozen oocyte pregnancy rate (56%) is equivalent to our frozen embryo pregnancy rate (45%). Patients, who have completed their families, find it easier to discard oocytes versus embryos.

Finally, women who make a personal choice to delay childbearing may be offered the option to preserve their oocytes with the potential for later use.

The two distinct techniques currently being used for oocyte cryopreservation are: 1) controlled-rate freezing and 2) vitrification. Controlled-rate freezing shares some similarities with the basic technology employed for embryo cryopreservation in nearly every IVF program. The technique involves the slow freezing of embryos in cryoprotectant solutions, often combined with a computer-controlled freezer to regulate temperature changes. Attempts to improve our understanding of oocyte cryobiology have been mostly empirical using trial and error. Only limited experience has been gained by adopting scientific models able to predict the effect of "cryo" stress imposed on oocytes using various freezing methods (Fuller and Paynter, 2004; Paynter, 2005). In the absence of properly designed studies, advances in clinical experience with oocyte freezing have been very limited. One of the major obstacles to the implementation of oocyte freezing had been the inability to achieve reproducible high survival rates owing to an important effect on the intracellular organelles. For example, due to its sensitivity at low temperature, the metaphase II spindle has always been considered susceptible to structural alterations which potentially might interfere with normal chromosome segregation at meiosis II. Additionally, the essential role of mitochondria in normal cell function, fertilization and early embryo development has previously been described (Jones et al., 2004).

Our recently developed modified freeze-thaw protocol has consistently shown high recovery rates, leading to optimism that oocyte storage could at last become available in clinical practice. But it remains to be demonstrated that excellent post-thaw survival coincides with cellular integrity and unaltered developmental competence. Therefore, prior to recommending the adoption of oocyte cryopreservation, one of our aims is to document the possible effect of cryo- preservation at the meiotic spindle and mitochondrial levels. An important aim of our study is to assess the post-thaw viability and organelle integrity of oocytes using: 1) a conservative technique [PolScope analysis of meiotic spindle] and 2) a non-conservative technique [Fluorescence microscopy analysis of the meiotic spindle and mitochondria] using our oocyte cryopreservation protocol.

Continuing development in freezing technology is occurring rapidly. It can be anticipated that in the near future, egg freezing will become as successful as embryo cryopreservation. Finally, as more clinical experience with egg freezing accumulates, acceptable outcome data will determine the future of egg freezing. Until then, oocyte cryopreservation should be used in carefully selected clinical cases with full disclosure to the patient regarding risks and limited success rates.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion into this study, each subject must satisfy the following criteria:

1. Participants must be aged 21 to 35 years
2. Body mass index (BMI) < 38.
3. Serum results for cycle day 3 FSH <10 mIU/ml.
4. Be willing and able to comply with the protocol for the duration of the study.
5. Have voluntarily provided written informed consent under WIRB, prior to any study-related procedure that is not part of normal medical care, with the understanding that the subjects may withdraw consent anytime without prejudice to their future medical care.
6. Have passed a psychological and physical screening.

Exclusion Criteria:

A patient may NOT be entered into the study if she presents with ANY of the following criteria:

1. Clinically significant systemic disease.
2. Known endometriosis Grade III - IV (ASRM classification).
3. Any previous cycle indicating a low response to gonadotropin stimulation (defined as retrieval of < 10 eggs at retrieval)
4. Previous ovarian surgery
5. Known allergy or hypersensitivity to recombinant gonadotropin preparations or any other study-related medications.
6. Known current substance abuse.
7. Simultaneous participation in another clinical trial.
8. Current smoker.
9. An extrauterine pregnancy within the last 3 months before OCP treatment commences.
10. Previous participation in similar study at different centers.

Ages: 21 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women of reproductive age who undergo controlled ovarian hyperstimulation (COH) for IVF are recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To document the freeze/thaw survival rates of human oocytes and to compare the structure changes in their meiotic spindle and mitochondria before and after cryopreservation. | When study complete

CONTACTS AND LOCATIONS:
Overall Officials: David G Diaz, MD, Principal Investigator — West Coast Fertility Centers
Locations (1):
- West Coast Fertility Centers, Fountain Valley, California, United States